CLINICAL TRIAL: NCT03679715
Title: Effects of the Montreal Museum of Fine Arts Participatory Art-based Activity on Health of Older Community Dwellers: THE A-HEALTH RCT STUDY
Brief Title: A-Health RCT: Effects of Participatory Art-based Activity on Health of Older Community Dwellers
Acronym: A-Health-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Principal Investigator, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-1493
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Social Interaction; Quality of Life; Health, Subjective
Keywords: Community-dwellers; older adults; museum; art

STUDY DESIGN:
Intervention Model Description: The design is a unicentre (Jewish General Hospital; Montreal, Quebec, Canada), clinical, randomized, controlled, single blinded (i.e.; investigators), superiority trial, with two parallel arms (Intervention and Control groups), comparative (comparison between Intervention and Control groups) and analyzed with the intention-to-treat.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants in the Intervention group will be participants of the museum participatory art-based activity.
  Interventions: Other: participatory art-based activity
- Control Group (No Intervention): The Control arm will be composed of older community dwellers matched on age and sex compared to the Intervention group but who will not be participants at the museum participatory art-based activity.

INTERVENTIONS:
Other: participatory art-based activity — The intervention is a participatory art-based activity which consists in making art in group, involving the participants directly in the creative process, allowing them to become co-authors of the work.
  In Montreal, Canada, participants will meet once per week for a 2h workshop from 2.00 PM to 4.00 PM at the MMFA in a dedicated room during a three month-period defining "a session". Two successive sessions will be setup; a winter and a spring sessions. Each session will be composed of 12 consecutive workshops.
  In Tokyo, Japan, participants will meet once per week for a 2h workshop at the Tokyo Fuji Museum in a dedicated room during a three month-period defining "a session". The session will be composed of 12 consecutive workshops.
  Arms: Intervention group

SUMMARY:
The overall objective of the study is to examine the effects of the Montreal Museum of Fine Arts (MMFA) participatory art-based activity on wellbeing, quality of life and health condition in older community dwellers.

Aging is often associated with worsening health and withdrawal from social activities, both increasing the risk of a poor quality of life. It has been reported that the practice of art, especially participatory art-based activity enhances wellbeing, quality of life and health condition of patients and older adults. Since October 2015, the Montreal Museum of Fine Arts (MMFA; Quebec, Canada) has successfully initiated a participatory art-based activity known as "Les Beaux-Jeudis" for older community dwellers living in Montreal. Recently, the investigator demonstrated that the MMFA participatory art-based activity improved wellbeing, quality of life and health condition of Montreal older community dwellers using a pre-post single arm, prospective and longitudinal design: it was not a randomized controlled trial (RCT) which is the gold standard to examine the effects of an intervention.

DETAILED DESCRIPTION:
Background. Recently, the investigator demonstrated that the Montreal Museum of Fine-Arts (MMFA) participatory art-based activity improved wellbeing, quality of life and health condition of Montreal older community dwellers using a pre-post single arm, prospective and longitudinal design. The main limitation of this pilot study was its design: it was not a randomized controlled trial (RCT) which is the gold standard to examine the effects of an intervention.

Objectives. The overall objective is to examine the effect of the MMFA participatory art-based activity on wellbeing, quality of life and health condition in older community dwellers.

The specific objectives are to compare the changes in 1) wellbeing, 2) quality of life and 3) health condition in older community dwellers participating in the museum participatory art-based activity (Intervention group) and in age and sex-matched older community dwellers who are not participants in the museum participatory art-based activity (Control group) during the same period of time. In addition, the compliance to museum participatory art-based activity in intervention will be examined. A second study, based on the same process, has been proceeded in Japan (Tokyo). With merging the 2 databases, we will study the impact of cultural specificities, comparing data collected in Montreal and data collected in Tokyo.

Methods. The design is a unicentre (Jewish General Hospital; Montreal, Quebec, Canada), clinical, randomized, controlled, single blinded (i.e.; investigators), superiority trial, with two parallel arms (Intervention and Control groups), comparative (comparison of Intervention and Control groups) and analyzed with the intention-to-treat.

The participants in the Intervention group will be participants of the museum participatory art-based activity. The Control group will be composed of older community dwellers matched on age and sex compared to the Intervention group but who will not be participate to the museum participatory art-based activity.

The follow-up period will be 3 months, which is the duration of a session of the museum participatory art-based activity. Assessment of wellbeing, quality of life and health condition will be performed at baseline, at the beginning of second and third months, and at the end of third month.

The same study has been developed and realized in Japan. Data collected in Canada will be merged with data collected in Japan and the analysis will be repeated for this international database.

ELIGIBILITY:
Inclusion Criteria:

1. Being 65 years and over
2. Having an Internet access with an electronic device (i.e.; laptop, computer, smartphone, tablet) at the participant's place of living as the repetitive assessments for this study will be performed on the web platform of the Centre of Excellence on Longevity of McGill University
3. Understanding and writing the language of the recruitment centre (i.e., French or English or Japanese)
4. Life expectancy estimated over 3 months as the duration of the follow-up is 3 months

Exclusion Criteria:

1. concomitant participation to another clinical trial,
2. having participated to a participatory art-based activity of the museums,
3. not speaking the language of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 235 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Health condition assessed by self-administered questionnaire (SAQ) | 3 months
  self-administered questionnaire (SAQ), score between 0 and 18, a higher score means a higher frailty

SECONDARY OUTCOMES:
Ability to use a computer assessed by Computer proficiency questionnaire self-questionnaire (CPQ) | 1 day
  Computer proficiency questionnaire self-questionnaire, self-estimation of different tasks on informatics devices quoted from Never tried to Very easily (high score for proficiency in informatics). Score for each categories is calculated from the mean of the sub-questions scored from 0 to 4
Well-being assessed by Warwick-Edinburgh Mental Well-being Scale self-questionnaire | 3 months
  Warwick-Edinburgh Mental Well-being Scale self-questionnaire, quoting statement of feelings and thought from None of the Time to All of the time, scoring from 14 to 70 (high score for a good well-being)
Quality of life of participants assessed by EuroQol-5D self-questionnaire | 3 months
  EuroQol-5D self-questionnaire, evaluating mobility, usual activities, self-care, pain, anxiety and mood, from No problem to Unable, scored from 5 to 25, High score meaning a bad quality of life
Compliance assessed counting the number of workshops completed during the 3-month period of intervention. | 3 months
  assessed counting the number of workshops completed during the 3-months period of intervention.
Satisfaction concerning the project assessed by self-questionnaire | 1 day
  self-questionnaire, qualitative (from 1 to 10: Dissatisfying to Satisfying), NO GLOBAL SCORE, each question is evaluated separately. A mean of all questions to have a global note (/10) will eventually be done for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (2):
- Jewish General Hospital, Montreal, Quebec, Canada
- Arts Alive, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cami M, Planta O, Matskiv J, Plonka A, Gros A, Beauchet O. Museum-based art activities to stay young at heart? Results of a randomized controlled trial. Front Med (Lausanne). 2024 Jan 5;10:1184040. doi: 10.3389/fmed.2023.1184040. eCollection 2023. PMID 38249982
- [Derived] Hayashi Y, Matskiv J, Galery K, Beauchet O. Productive arts engagement at the Tokyo Fuji Art Museum and its health effects on the older Japanese population: results of a randomized controlled trial. Front Med (Lausanne). 2023 Jul 6;10:1188780. doi: 10.3389/fmed.2023.1188780. eCollection 2023. PMID 37484855
- [Derived] Beauchet O, Cooper-Brown LA, Hayashi Y, Deveault M, Launay CP. Improving the mental and physical health of older community-dwellers with a museum participatory art-based activity: results of a multicentre randomized controlled trial. Aging Clin Exp Res. 2022 Jul;34(7):1645-1654. doi: 10.1007/s40520-022-02139-3. Epub 2022 May 17. PMID 35578103
- [Derived] Beauchet O, Cooper-Brown L, Hayashi Y, Galery K, Vilcocq C, Bastien T. Effects of "Thursdays at the Museum" at the Montreal Museum of Fine Arts on the mental and physical health of older community dwellers: the art-health randomized clinical trial protocol. Trials. 2020 Aug 12;21(1):709. doi: 10.1186/s13063-020-04625-3. PMID 32787893